CLINICAL TRIAL: NCT00280137
Title: Health-related Quality of Life Measure in Pediatric Lupus
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Hospital for Special Surgery, New York (Other); St. Barnabas Medical Center (Other); Hackensack Meridian Health (Other); University of Chicago (Other); The Cleveland Clinic (Other); Children's Hospital Los Angeles (Other); Legacy Health System (Other); University Hospitals Cleveland Medical Center (Other); Tufts Medical Center (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0220044879
Record Dates: First submitted 2006-01-13; First posted 2006-01-20 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Systemic Lupus Erythematosus; Quality of Life
Keywords: Quality of Life; Pediatric Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the psychometric properties of a brief quality of life (QOL) instrument for use in pediatric systemic lupus erythematosus (SLE). The purpose of this prospective study is primarily to determine the validity and reliability of a new health-related quality of life (HRQOL) measure in children with systemic lupus erythematous (SLE). We wish to secondarily examine concordance between child- and parent-reports of the HRQOL measure and identify factors associated with poorer HRQOL in them.

Earlier studies have shown that SLE significantly impacts QOL in adults. At present, there is no disease-specific instrument for measuring HRQOL in children with SLE. In response to these concerns, we developed the "Simple Measure of Impact of Lupus Erythematosus in Youngsters© (SMILEY©). Establishing the validity and reliability of SMILEY©, examining child-parent agreement and identifying factors associated with poorer HRQOL will enable us to measure the impact of SLE in children, and formulate appropriate interventions for this sensitive population. We plan the following specific aims:

1. to determine construct validity and reliability of SMILEY© child and parent versions in children with SLE using gold standards (Pediatric Quality of Life inventory - PedsQL generic and rheumatology modules, Childhood Health Assessment Questionnaire -CHAQ)
2. to determine responsiveness of SMILEY©
3. to examine level of agreement between child- and parent-reports of SMILEY© in children with SLE
4. to identify medical (steroid use, use of disease modifying agents such as cytoxan, cellcept, thalidomide, or cyclosporine, disease duration, disease activity and disease damage etc.) and psychosocial (self-concept, socioeconomic status) factors that affect HRQOL (as measured by child- and parent-reports of SMILEY© and PedsQL generic and rheumatology modules) and physical function 5) to translate, adapt and validate SMILEY in different languages

DETAILED DESCRIPTION:
Pediatric lupus is a chronic multisystem rheumatic disease, associated with significant medical and psychosocial implications. Frequent physician visits for routine, urgent or emergent care, limitation of activities, medication side effects, change in body image, fear of the future, and missing school are all disruptive to the patients and parents and impact all spheres of their lives. There is no lupus-specific questionnaire designed to measure the well-being of children with this disease. We developed a brief questionnaire, "Simple Measure of Impact of Lupus Erythematosus in Youngsters© (SMILEY©) with both child and parent versions. We conducted further research about how children/parents feel about having/their children having lupus and used those responses to modify the preliminary SMILEY©. After several iterations, the SMILEY with 26 questions was developed with parallel child- and parent-versions with responses in the form of 5 faces-scale denoting different expressions, in order to ensure easy comprehension across different ages and cultures.

During their visit, information about their lupus will be collected from the children and parents, and they will be asked to complete the SMILEY© and questionnaires measuring quality of life, physical function, self-esteem and behavior. They will be given an additional copy of SMILEY©, which they will be asked to complete within 10 days of their initial evaluation and return by mail (self-addressed, stamped envelope will be provided). Then both children and legal guardians will again be asked to complete questionnaires including SMILEY© during their subsequent visits at least every 3-6 month intervals or earlier if there has been a change in disease activity as determined by the physician. Medication use, disease activity and disease severity assessments will be made by the physician with initial and subsequent evaluations. We will determine the psychometrics properties of SMILEY and responsiveness to change in disease activity.

Both national and international sites will be included in the study. SMILEY in addition will be translated and adapated to different languages and subsequently validated. This study will provide valuable information about the impact of lupus on their overall well-being. Being a brief, valid, reliable and easy to administer instrument, SMILEY© would be suitable for use across different age groups, languages and cultures. SMILEY© will be used as an important clinical outcome tool in both clinical and research arenas, thus enabling us to formulate appropriate interventions.

ELIGIBILITY:
Inclusion Criteria:

* (1) Willing to participate
* (2) Have a child with SLE that meets eligibility criteria for the study

Exclusion Criteria:

* (1) Subjects who are not well enough to complete the questionnaires
* (2) Physical or mental disabilities which would seriously affect the individual's ability to understand the informed consent or study questionnaires
* (3) Refusal to participate

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population will consist of outpatients during clinics visits and inpatients during hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2004-06; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life - scores of the SMILEY scale for child and parent reports | At different points of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi N Moorthy, MD, MS, Principal Investigator — UMDNJ/RWJUH Department of Pediatrics
Locations (11):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - La Rabida Children's Hospital - The University of Chicago, Chicago, Illinois
  - New England Medical Center -Tufts, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - University of Medicine and Dentistry - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York
  - The CLeveland CLinic, Cleveland, Ohio
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Legacy Health System, Portland, Oregon

REFERENCES:
- [Background] Moorthy LN, Robbins L, Harrison MJ, Peterson MG, Cox N, Onel KB, Lehman TJ. Quality of life in paediatric lupus. Lupus. 2004;13(4):234-40. doi: 10.1191/0961203304lu1003oa. PMID 15176658
- [Background] Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH. Derivation of the SLEDAI. A disease activity index for lupus patients. The Committee on Prognosis Studies in SLE. Arthritis Rheum. 1992 Jun;35(6):630-40. doi: 10.1002/art.1780350606. PMID 1599520
- [Background] Stoll T, Stucki G, Malik J, Pyke S, Isenberg DA. Association of the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index with measures of disease activity and health status in patients with systemic lupus erythematosus. J Rheumatol. 1997 Feb;24(2):309-13. PMID 9034988
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Singh G, Athreya BH, Fries JF, Goldsmith DP. Measurement of health status in children with juvenile rheumatoid arthritis. Arthritis Rheum. 1994 Dec;37(12):1761-9. doi: 10.1002/art.1780371209. PMID 7986222